CLINICAL TRIAL: NCT03736889
Title: A Single-Arm, Multi-Center, Open-Label, Phase 2 Study to Evaluate Efficacy and Safety of Tislelizumab (BGB-A317), an Anti-PD-1 Monoclonal Antibody, as Monotherapy in Patients With Previously-Treated Locally Advanced Unresectable or Metastatic Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) Solid Tumors
Brief Title: Tislelizumab (Anti-Programmed Cell Death Protein-1 (PD-1) Antibody) in MSI-H or dMMR Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-209; CTR20180867 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2018-10-31; First posted 2018-11-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: MSI-H/dMMR Solid Tumors
Keywords: MSI-H/dMMR; Solid tumors; PD-1
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab (BGB-A317) Injection (Experimental)
  Interventions: Drug: Tislelizumab (BGB-A317)

INTERVENTIONS:
Drug: Tislelizumab (BGB-A317) — Anti-PD-1 Antibody

SUMMARY:
In this Phase 2, Single-Arm, Multi-Center, Open-Label Study, participants with previously treated locally advanced unresectable or metastatic solid tumors with mismatched repair deficient (dMMR) or microsatellite instability-high (MSI-H) will be treated with anti-PD-1 Monoclonal Antibody Tislelizumab (BGB-A317).

ELIGIBILITY:
Key Inclusion Criteria:

1. Having histological confirmed diagnosis of malignancy
2. Having locally advanced unresectable or metastatic solid tumors with MSI-H or dMMR
3. Having received prior cancer therapy regimen(s) for advanced disease.
4. At least 1 measurable lesion as defined per RECIST Version (v) 1.1
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
6. Adequate organ function

Key Exclusion Criteria:

1. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
2. Active leptomeningeal disease or uncontrolled brain metastasis.
3. Clinically significant pleural effusion, pericardial effusion or ascites
4. Active autoimmune diseases or history of autoimmune diseases that may relapse
5. Any active malignancy
6. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug
7. Having a history of interstitial lung disease, non-infectious pneumonitis, pulmonary fibrosis, acute lung diseases, or uncontrolled systemic diseases (including but not limited to diabetes, hypertension, etc.)
8. Participants with uncontrolled diabetes or uncontrolled electrolyte disorders despite standard medical management
9. Having severe chronic or active infections
10. A known history of human immunodeficiency virus infection
11. Child - Pugh B or greater cirrhosis
12. Any major surgical procedure ≤ 28 days before the first dose of study drug
13. Prior allogeneic stem cell transplantation or organ transplantation

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate assessed by Independent Review Committee per Response Evaluation Criteria in Solid Tumors Version 1.1 | Up to 2 years

SECONDARY OUTCOMES:
Duration of response assessed by Independent Review Committee and by investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | Up to 2 years
Time to response assessed by Independent Review Committee and by investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | Up to 2 years
Progression-free survival assessed by Independent Review Committee and by investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | Up to 2 years
Disease control rate assessed by Independent Review Committee and by investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | Up to 2 years
Overall survival | Up to 2 years
Objective response rate assessed by investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | Up to 2 years
Safety and tolerability assessment per the number of participants experiencing Treatment-Emergent Adverse Event (TEAE) as assessed by CTCAE v5.0 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (29):
- China (29):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Affiliated Hospital of Military Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - Huizhou First Hospital, Huizhou, Guangdong
  - Meizhou People Hospital, Meizhou, Guangdong
  - The Peoples Hospital of Hechi, Hechi, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The General Hospital of Shenyang Military, Shenyang, Liaoning
  - Yidu Central Hospital of Weifang, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The First Peoples Hospital of Yibin, Yibin, Sichuan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang